CLINICAL TRIAL: NCT00725140
Title: Standardized sTudy With Almotriptan in eaRly Treatment of Migraine, START. An International, Open-label, Single Arm, Effectiveness and Safety Study of Almotriptan in Primary Care Setting
Brief Title: Standardized sTudy With Almotriptan in eaRly Treatment of Migraine
Acronym: START
Status: Completed | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: M/31416/51; EudraCT: 2007-003392-39; Spanish AEM: ALM-ALM-2008-01
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Migraine
Keywords: Migraine; Early intervention; Primary Care; Almotriptan
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single

SUMMARY:
This is a observational, open, prospective, single arm cohort study within authorized SPC conditions to describe the effectiveness of Almotriptan in treating acute migraine attacks when pain is mild and in the first hour of pain in everyday primary care clinical practice.

DETAILED DESCRIPTION:
Primary Objective:

To describe the effectiveness of Almotriptan in treating acute migraine attacks when pain is mild and in the first hour of pain in everyday primary care clinical practice.

Secondary Objectives:

1. Influence of an educational intervention on the early intake of the treatment
2. Influence of medication history or concomitant medication on treatment results
3. Influence of migraine triggers on treatment results
4. Influence of stress on treatment results
5. Tolerability profile validation
6. Patients' satisfaction
7. Reasons for delaying migraine treatment intake

ELIGIBILITY:
Inclusion Criteria:

1. History of a confirmed diagnosis of migraine that meets the IHS diagnosis criteria of migraine with or without aura for at least one year.
2. Patients with a history of migraine headaches progressing from mild to at least moderate pain intensity if untreated on a scale of no pain (0), mild (1), moderate (2), or severe (3) within the past year.
3. Migraine headache frequency of 2 to 6 per month for the past 3 months.
4. Male or female aged 18 to 65 years.
5. Able to differentiate a migraine headache from an interval (e.g., tension-type) headache.

8.Female patients of childbearing potential must not suspect to be pregnant and have an effective method of birth control for at least 30 days prior to study entry and throughout the study.

11.After full explanation, patients must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study.

12.Patients must either use Almotriptan for their migraine acute attacks treatment or prove through the ANAES scale in the basal visit that a change in their treatment approach is required.

Exclusion Criteria:

1. Patients, who in the opinion of the investigator, should not be enrolled in the study because of the precautions, warnings or contraindications sections of the Almotriptan Summary of Product Characteristics.
2. Patients who have had 15 or more headache days per month in the previous 6 months (chronic daily headache), or patients having a migraine headache frequency of more than 6 per month for the past 3 months.
3. Patients with onset of migraine after age 50.
4. Patients who routinely experience any other type of headache that would confound discrimination from a migraine.
5. Patients who have exclusively migraine aura without headache.
6. Patients who typically experience vomiting with their headaches.
7. Patients with hemiplegic or basilar type migraines.
8. Patients who typically have headaches that occur predominantly upon awakening in the morning.
9. Patients who have previously discontinued Almotriptan therapy due to an adverse event or lack of efficacy.

11.Patients taking any of the prohibited concomitant medications listed in Section 10.3.1 of the protocol.

12.Patients who have used any of the following medications within 7 days of study entry and during the trial: sustained release opioids and/or semi-synthetic or long acting opioids.

16.Women who are pregnant or lactating.

18.Patients who have received an investigational drug or used an investigational device within 30 days of study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Following SPC conditions and study requirements, male or female of 18 to 65 years old with a minimum of one year of migraine history (International Headache Society criteria, see criteria attached in the protocol Annex 1) of moderate or severe intensity and with a frequency of 2 to 6 attacks per month for the past 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pain Free | 2 h from intake

SECONDARY OUTCOMES:
Sustained Pain Free | 24 h
SNAE (Sustained pain free and No Adverse Events) | 24 h
Relapse | 24 h
Second tablet / rescue medication use | 24 h
Associated symptoms presence evolution: Nausea, Vomiting, Photophobia, Phonophobia. | Basal - 2h - 24h
Migraine attack duration | 24 h
Time loss (functional disability) | 24 h
Patients' satisfaction: | Basal - After each attack
Adverse Events | From recruitment to study end or AE resolution
Consistency of response to treatment between attacks (2 h PF in 2/3 attacks) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel Lanteri-Minet, Dr, Study Chair — Pain Evaluation and Treatment Department, Hopital Pasteur, Nice, France
Locations (3):
- 28 GPs across France, Diverse, France
- 26 GPs across Italy, Diverse, Italy
- 26 GP practices across Spain, Diverse, Spain

REFERENCES:
- [Derived] Lanteri-Minet M, Diaz-Insa S, Leone M, Vila C, Clissold SP; START Study. Efficacy of almotriptan in early intervention for treatment of acute migraine in a primary care setting: the START study. Int J Clin Pract. 2010 Jun;64(7):936-43. doi: 10.1111/j.1742-1241.2010.02379.x. PMID 20584227